CLINICAL TRIAL: NCT03741127
Title: Open Label, Multicenter, Long-Term Follow-Up Study for Subjects Treated With P-BCMA-101
Brief Title: Long-Term Follow-Up Study for Subjects Treated With P-BCMA-101
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Poseida Therapeutics, Inc. (Industry)
Collaborators: California Institute for Regenerative Medicine (CIRM) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: P-BCMA-101-002
Record Dates: First submitted 2018-11-07; First posted 2018-11-14 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-01

CONDITIONS: Multiple Myeloma
Keywords: CAR-T cells
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- P-BCMA-101 treated (Other): Patients who received previous treatment with P-BCMA-101. Rimiducid may be administered as indicated.
  Interventions: Drug: Rimiducid may be administered as indicated

INTERVENTIONS:
Drug: Rimiducid may be administered as indicated — Patients who received P-BCMA-101 in a previous trial will be evaluated in this trial for long term safety and efficacy. Rimiducid (safety switch activator) may be administered as indicated.
  Other Names: Rimiducid (safety switch activator)

SUMMARY:
Subjects are enrolled in this study following completion or early discontinuation from a Poseida sponsored or supported study of P-BCMA-101 T cells and will be followed for a total of 15 years post treatment from the last P-BCMA-101 treatment. Subjects will be monitored for safety and efficacy to assess the risk of delayed adverse events (AEs) and assess long-term efficacy, and PK and quantification of P-BCMA-101 T cells. Rimiducid may be administered as indicated.

DETAILED DESCRIPTION:
Per Health Authorities guidelines for gene therapy medicinal products that utilize integrating vectors (FDA, 2006; Guidance for Industry, Gene Therapy Clinical Trials-Observing Subjects for Delayed Adverse Events), long term safety and efficacy follow up of treated subjects is required. Subjects are enrolled in this study following completion or early discontinuation from a Poseida sponsored or supported study of P-BCMA-101 T cells and will be followed for a total of 15 years post treatment from the last P-BCMA-101 treatment. Subjects will be monitored for safety and efficacy to assess the risk of delayed adverse events (AEs) and assess long-term efficacy, and PK and quantification of P-BCMA-101 T cells. Rimiducid may be administered as indicated.

Study visits Subjects will only enter this protocol after completing or discontinuing from their primary P-BCMA-101 protocol.

Once enrolled in this protocol a subject will return for regular follow-up depending on when they last received P-BCMA-101 on their primary protocol:

* Every 3 months until the end of the first year after P-BCMA-101 treatment
* Every 6 months until the end of the third year after P-BCMA-101 treatment
* Then yearly until the end of the 15th year after P-BCMA-101 treatment (ie. if a subject discontinues from their primary protocol 2 years after receiving P-BCMA-101, they will be entering this study at the beginning of the 3rd year, and will remain on this study for 13 years).

Subjects will undergo serial assessment of safety, chemistry, hematology, and disease response as specified in the Schedule of Events. Subjects will further undergo a physical exam and medical history, and anti-myeloma medications, related AEs, new malignancies, new or exacerbated clinically significant neurologic, hematologic, rheumatologic or other autoimmune disorders will be recorded. After progressive disease (PD) has been confirmed for a subject after P-BCMA-101 administration, visits may be performed remotely (AEs collected by telephone and laboratory studies completed at a local facility).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have received P-BCMA-101 and completed or discontinued early from a Poseida sponsored treatment protocol.
* Subject has provided informed consent.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-10-29 (Actual); Primary Completion 2032-08 (Estimated); Study Completion 2032-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Treatment with P-BCMA-101 through year 15
  Incidence and severity of treatment-emergent adverse events to evaluate the long-term safety of P-BCMA-101

SECONDARY OUTCOMES:
Anti-myeloma effect of P-BCMA-101 (Response Rate) | Treatment with P-BCMA-101 through year 15
  Percentage of patients with complete response (CR), very good partial response (VGPR), or partial response (PR) according to the International Myeloma Working Group (IMWG) Uniform Response Criteria for Multiple Myeloma
Anti-myeloma effect of P-BCMA-101 (Time to Response) | Treatment with P-BCMA-101 through year 15
  Time from P-BCMA-101 administration to time of first documented response (PR or better) according to the International Myeloma Working Group (IMWG) Uniform Response Criteria for Multiple Myeloma.
Anti-myeloma effect of P-BCMA-101 (Duration of Response) | Treatment with P-BCMA-101 through year 15
  Time from complete response (CR), very good partial response (VGPR), or partial response (PR) to progressive disease according to the International Myeloma Working Group (IMWG) Uniform Response Criteria for Multiple Myeloma.
Anti-myeloma effect of P-BCMA-101 (Progression Free Survival) | Treatment with P-BCMA-101 through year 15
  Time from P-BCMA-101 treatment to progressive disease according to the International Myeloma Working Group (IMWG) Uniform Response Criteria for Multiple Myeloma, or death
Anti-myeloma effect of P-BCMA-101 (Overall Survival) | Treatment with P-BCMA-101 through year 15
  Duration of survival from time of treatment with P-BCMA-101
Concentration of P-BCMA-101 cells | Treatment with P-BCMA-101 through year 15
  Concentration of P-BCMA-101 cells in blood and bone marrow over time
Biomarkers for P-BCMA-101 (BCMA Cells) | Treatment with P-BCMA-101 through year 15
  The persistence of anti-tumor effect of P-BCMA-101 and its relationship to persistence of P-BCMA-101 cells, BCMA tumor surface expression and circulating BCMA.
Biomarkers for P-BCMA-101 (Cell Count) | Treatment with P-BCMA-101 through year 15
  Absolute B and T lymphocyte count
Biomarkers for P-BCMA-101 (Expansion) | Treatment with P-BCMA-101 through year 15
  Expansion and/or persistence of P-BCMA-101 T cells
Incidence of adverse events related to rimiducid, if indicated | Rimiducid infusion through Year 15 after P-BCMA-101 infusion, if applicable
  Incidence of adverse events related to rimiducid, if indicated
Effect of rimiducid on grade of P-BCMA-101-related adverse events | Rimiducid infusion through Year 15 after P-BCMA-101 infusion, if applicable
  Effect of rimiducid on grade of P-BCMA-101-related adverse events as assessed by CTCAE v4.03, if indicated.

CONTACTS AND LOCATIONS:
Overall Officials: Semira Sheikh,, M.D., P.h.D, Study Director — Sponsor Medical Director
Locations (13):
- United States (13):
  - University of California Davis, Davis, California
  - University of California, San Diego, San Diego, California
  - University of California San Francisco, San Francisco, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - University of Chicago, Chicago, Illinois
  - University of Kansas Cancer Center, Westwood, Kansas
  - University of Maryland Greenebaum Comprehensive Cancer Center, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Wayne State - Karmanos Cancer Institute, Detroit, Michigan
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute at Tennessee Oncology, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No